CLINICAL TRIAL: NCT02764398
Title: Prospective Analysis of Serious Cardio-respiratory Events During Ophthalmic Artery Chemotherapy for Retinoblastoma Under a Deep and Standardized Anesthesia
Brief Title: Cardio-respiratory Events During Ophthalmic Artery Chemotherapy for Retinoblastoma Under a Deep Anesthesia
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_2016_1
Record Dates: First submitted 2016-05-01; First posted 2016-05-06 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Background: Serious adverse cardio-respiratory events (SCRE) occur during super selective ophthalmic artery chemotherapy for retinoblastoma in children. SCRE mechanism remains unclear but may be attributed to an autonomic nervous reflex induced by catheterization of the ophthalmic artery. The investigators hypothesize that inadequacy between depth of anesthesia and catheter stimulation might be a support cause of these SCRE.

Methods: Children requiring super selective ophthalmic artery chemotherapy for retinoblastoma are prospectively included in this observational study. Endovascular procedures are performed under standardized and deep general anesthesia with sevoflurane, sufentanil and rocuronium. SCRE are strictly pre-defined and included arterial hypotension, bradycardia and bronchospasm. SCRE are recorded and the factors influencing their occurrence are investigated.

ELIGIBILITY:
Inclusion Criteria:

* superselective ophthalmic artery chemotherapy for retinoblastoma required

Exclusion Criteria:

* no

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children requiring superselective ophthalmic artery chemotherapy for retinoblastoma
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Serious adverse cardio-respiratory events during ophthalmic artery chemotherapy for retinoblastoma. | from the beginning of general anesthesia until the end of injection of chemotherapy in the ophthalmic artery, assessed up to 120 minutes.